CLINICAL TRIAL: NCT05218655
Title: An Open-Label, Safety Study for Previously Treated Vatiquinone (PTC743) Subjects With Inherited Mitochondrial Disease
Brief Title: A Safety Study for Previously Treated Vatiquinone (PTC743) Participants With Inherited Mitochondrial Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC743-CNS-005-LSEP; 2022-000375-39 (EudraCT Number)
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Results first posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Inherited Mitochondrial Disease
Keywords: Leigh syndrome; Alpers Syndrome; mitochondrial encephalomyopathy; MELAS; MERRF; PCH6; refractory epilepsy
MeSH Terms: conditions — Leigh Disease; Diffuse Cerebral Sclerosis of Schilder; Mitochondrial Encephalomyopathies; MELAS Syndrome; MERRF Syndrome; Drug Resistant Epilepsy | interventions — alpha-tocotrienol quinone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vatiquinone (Experimental): Participants will receive vatiquinone oral solution (100 milligrams [mg]/milliliter [mL]), up to 400 mg, administered orally or via feeding tube 3 times daily (TID).
  Interventions: Drug: Vatiquinone

INTERVENTIONS:
Drug: Vatiquinone — Vatiquinone will be administered per dose and schedule specified in the arm description.
  Other Names: PTC743

SUMMARY:
The primary objective of this study is to assess the safety of vatiquinone in participants with inherited mitochondrial disease who had prior exposure to vatiquinone in a PTC/BioElectron sponsored (previously Edison) clinical study or treatment plan.

The study will continue until vatiquinone becomes commercially available or the program is terminated.

ELIGIBILITY:
Inclusion Criteria:

* Participants with inherited mitochondrial disease including Leigh syndrome, Alpers syndrome, mitochondrial encephalomyopathy, lactic acidosis and stroke-like episodes (MELAS), myoclonic epilepsy with ragged-red fibers (MERRF), pontocerebellar hypoplasia type 6 (PCH6), or other mitochondrial disease who participated in a previous vatiquinone clinical study or treatment plan.
* Women of childbearing potential must have a negative pregnancy test at screening/baseline and agree to abstinence or the use of at least 1 of the highly effective forms of contraception as specified in the protocol (with a failure rate of <1% per year when used consistently and correctly). Highly effective contraception or abstinence must be continued for the duration of the study, and for up to 30 days after the last dose of study drug.
* Fertile men who are sexually active with women of childbearing potential and who have not had a vasectomy, must agree to use a barrier method of birth control during the study and for up to 30 days after the last dose of study drug.

Exclusion Criteria:

* Current participation in any other interventional study.
* Pregnancy or breast feeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Penematsa, MD, Study Director — PTC Therapeutics
Locations (26):
- United States (14):
  - University of California, San Diego Altman Clinical and Translational Research Institute, La Jolla, California
  - Stanford University, Stanford, California
  - Yale Medicine, New Haven, Connecticut
  - Children's National, Washington D.C., District of Columbia
  - Child Neurology Center of Northwest Florida, Gulf Breeze, Florida
  - The Johns Hopkins University, Baltimore, Maryland
  - Columbia University Medical Center - CUMC, New York, New York
  - Akron Children's Hospital, Akron, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital of Philadelphia - CHOP, Philadelphia, Pennsylvania
  - Medical University of South Carolina - MUSC, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - UT Health The University of Texas, Houston, Texas
  - Seattle Children Hospital, Seattle, Washington
- France (4):
  - Chu Angers, Angers
  - CHU Montpellier - Hopital Saint-Eloi, Montpellier
  - Hopital Necker-Enfants Malades, Paris
  - Hôpital de Hautepierre - Hôpitaux Universitaires de Strasbourg, Strasbourg
- Ospedale Pediatrico Bambino Gesù, Roma, Italy
- PTC Clinical Site, Japanese City, Japan
- Instytut Pomnik - Centrum Zdrowia Dziecka, Warsaw, Poland
- Spain (3):
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Ruber Internacional, Madrid
- United Kingdom (2):
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 103 participants were screened, of which 101 participants were enrolled in the study and received at least 1 dose of vatiquinone.
Groups:
- Vatiquinone: Participants received vatiquinone oral solution (100 milligrams [mg]/milliliter [mL]), up to 400 mg, administered orally or via feeding tube 3 times daily (TID).
Period: Overall Study
Arm/Group | Vatiquinone
Started | 101
Received At Least 1 Dose of Study Drug | 101
Completed | 0
Not Completed | 101
Not completed — Adverse Event | 6
Not completed — Sponsor's decision | 85
Not completed — Death | 1
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 3
Not completed — Other than specified | 3

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of vatiquinone in the study.
Arm/Group | Vatiquinone
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.5 (11.56) [lower limit 11.56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian/Alaska Native | 1
  Race: Asian | 8
  Race: Black/African American | 2
  Race: White | 83
  Race: Other | 1
  Race: Unknown | 1
  Race: Missing | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 9
  Ethnicity: Not Hispanic or Latino | 86
  Ethnicity: Not Reported | 3
  Ethnicity: Unknown | 2
  Ethnicity: Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AEs included both serious adverse events (SAEs) and non-serious AEs. A TEAE was defined as an AE that had an onset date or date of worsening on or after the first dose of study drug and within 30 days of the date of the last dose of treatment. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: Baseline (Day 1) up to 30 days after last dose of study drug (956 days)
Population: Safety population included all participants who received at least 1 dose of vatiquinone in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Vatiquinone
Number analyzed (Participants) | 101
Participants | 91

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to 30 days after last dose of study drug (956 days)
Description: Safety population included all participants who received at least 1 dose of vatiquinone in the study.
Groups:
- Vatiquinone: Participants received vatiquinone oral solution (100 mg/mL), up to 400 mg, administered orally or via feeding tube TID.
Arm/Group | Vatiquinone
All-Cause Mortality (participants affected / at risk) | 7/101
Serious Adverse Events (participants affected / at risk) | 45/101
Other Adverse Events (participants affected / at risk) | 59/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vatiquinone (N=101)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (2)
Fanconi syndrome (Congenital, familial and genetic disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (2)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Death (General disorders) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Generalised oedema (General disorders) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
COVID-19 (Infections and infestations) | 3 (3)
Influenza (Infections and infestations) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 10 (11)
Pneumonia aspiration (Infections and infestations) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2)
Rhinovirus infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Streptococcal infection (Infections and infestations) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Urosepsis (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Mitochondrial cytopathy (Metabolism and nutrition disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1)
Change in seizure presentation (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 2 (2)
Myoclonus (Nervous system disorders) | 1 (1)
Optic neuritis (Nervous system disorders) | 1 (2)
Seizure (Nervous system disorders) | 2 (3)
Status epilepticus (Nervous system disorders) | 3 (4)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 (16)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary amyloidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tracheostomy (Surgical and medical procedures) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vatiquinone (N=101)
Diarrhoea (Gastrointestinal disorders) | 6 (7)
Vomiting (Gastrointestinal disorders) | 11 (15)
Pyrexia (General disorders) | 12 (24)
COVID-19 (Infections and infestations) | 13 (14)
Nasopharyngitis (Infections and infestations) | 7 (9)
Pneumonia (Infections and infestations) | 6 (9)
Respiratory tract infection (Infections and infestations) | 6 (10)
Upper respiratory tract infection (Infections and infestations) | 14 (19)
Urinary tract infection (Infections and infestations) | 9 (9)
Gamma-glutamyltransferase increased (Investigations) | 6 (7)
Seizure (Nervous system disorders) | 9 (9)

LIMITATIONS AND CAVEATS:
The study was terminated early as PTC discontinued clinical development of vatiquinone for this indication based on prior clinical study results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the Sponsor for review. The Sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT05218655/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT05218655/SAP_001.pdf